CLINICAL TRIAL: NCT06705530
Title: An Interventional Open-label, Single-group, Phase I/II Study to Evaluate the Tolerability, Safety, and Efficacy of an Anti-CD19 CAR-T Product in Adult Patients With Relapsed or Refractory Forms of B-cell Lymphoproliferative Disorders
Brief Title: A Study to Evaluate the Tolerability, Safety, and Efficacy of an Anti-CD19 CAR-T Product in Patients With B-cell Lymphoproliferative Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HemC101-01-01
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-Hodgkin Lymphoma, B-cell; Acute Lymphoblastic Leukemia ALL
Keywords: CAR-T; B-cell lymphoma; non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hem101 Arm (Experimental): The investigational product (Hem101) will be administered as an intravenous infusion twice to each patient, on Day 1 and Day 2 of the dose if the first dose is well tolerated
  Interventions: Biological: Hem101

INTERVENTIONS:
Biological: Hem101 — CAR-T lymphocytes specific to CD19 B-cell antigen
  Other Names: Hemagenleukleucel

SUMMARY:
This study is testing a new type of treatment called anti-CD19 CAR-T cell therapy for adults with certain blood cancers that have returned or did not respond to previous treatments. CAR-T cells are a type of immune cell that is specially designed in a lab to target and destroy cancer cells with a marker called CD19. The main goals of this study are to find out if this treatment is safe, how well patients tolerate it, and how effective it is at controlling cancer.

The study will include 60 adults, ages 18-70, who meet specific criteria for participation. Patients will first receive a short course of chemotherapy to prepare their bodies for the CAR-T cells. The CAR-T cells will then be given in two doses through an IV. Patients will be monitored closely in the hospital for about a month to check for any side effects and see how their cancer responds. The researchers will also follow up with patients over time to learn more about how long the CAR-T cells stay active, how well they fight cancer, and the overall health of the patients after treatment.

DETAILED DESCRIPTION:
This Phase I/II open-label, single-arm clinical trial evaluates the safety, tolerability, and efficacy of anti-CD19 CAR-T cell therapy in adult patients with relapsed or refractory B-cell lymphoproliferative disorders, including B-cell acute lymphoblastic leukemia (B-ALL) and non-Hodgkin lymphoma (NHL). Anti-CD19 CAR-T therapy uses genetically modified T cells engineered to recognize and destroy cancer cells with the CD19 antigen. The investigational therapy utilizes second-generation CAR-T cells. The primary objective of the study is to assess the overall response rate (ORR) at Day 28. In contrast, secondary objectives include evaluating progression-free survival (PFS), duration of response (DoR), and overall survival (OS).

The trial will recruit 60 participants between 18 and 70 years old who meet specific eligibility criteria, including CD19 expression on tumor cells and adequate organ function. Participants will first undergo lymphodepletion to prepare their immune systems for CAR-T cell infusion. The CAR-T therapy will be administered in two doses via intravenous infusion. This dosing regimen is designed to optimize safety and maximize therapeutic benefit. The treatment period includes close inpatient monitoring for at least 14 days, followed by additional outpatient assessments.

Safety and tolerability are key components of the study, with close observation for potential side effects such as cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS). Other safety measures include evaluating organ function, monitoring for infections, and assessing the presence of antibodies against CAR-T cells. Efficacy will be determined based on tumor responses, measured as complete or partial remission, and by tracking the persistence and expansion of CAR-T cells in the blood.

This study is being conducted at a single clinical center in Russia and is sponsored by the National Medical Research Center of Hematology, Ministry of Health of Russia. The expected duration for each participant is approximately 53 days, with long-term follow-up planned to evaluate the durability of treatment responses and overall survival outcomes. The findings from this study will help determine whether anti-CD19 CAR-T therapy is a viable treatment option for patients with difficult-to-treat B-cell blood cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with B-cell lymphoproliferative disorders:

1a. In cases of B-cell lymphoproliferative disorders developed from lymphocyte precursors (ALL/LBL), the disease status satisfies one of the following criteria:

* Failure of induction (primary-refractory course or MOB persistence), absence of clinical and hematologic remission after first-line therapy,
* MOB persistence with achieved second and subsequent clinical and morphologic remissions,
* Early medullary or combined relapse if the duration of the first remission is not more than 12 months, provided the disease is stabilized,
* Confirmed MOB relapse,
* Second and subsequent relapses, including neurorelapse,
* Refractory disease course after two or more lines of chemotherapy,
* Relapsed or refractory disease after allo-HSCT with transplantation performed more than 100 days ago and more than 4 weeks after withdrawal of immunosuppressive therapy before inclusion.

  1. b. In the case of Ph-positive ALL/LBL:
* Molecular relapse, advanced relapse, isolated neurorelapse, or refractory disease after the use of more than 2 lines of ITC.

  1c. In cases of aggressive B-cell non-Hodgkin's lymphoma, disease status satisfies one of the following criteria:
* Absence of remission after 1-2 courses of intensive chemotherapy or in the presence of factors of unfavorable prognosis (TP53 mutation, co-expression of c-MYC and BCL2, abnormalities of c-MYC, BCL2, BCL6, and other genes),
* Disease progression on chemotherapy in the form of the appearance of a new lesion focus or increase of the initial focus by at least 50% during therapy,
* Relapse within 12-18 months after the end of chemotherapy, regardless of the presence or absence of factors of unfavorable prognosis,
* Resistance to 2 or more prior lines of therapy.

  1d. In cases of indolent B-cell non-Hodgkin's lymphoma, disease status satisfies one of the following criteria:
* early relapse (POD 24) in patients with contraindications to auto-HSCT,
* absence of clinical and hematologic remission after 1 line of therapy in the presence of TR53 mutation,
* relapse in the presence of signs of transformation into aggressive lymphoma,
* resistance to the previously performed 2 or more lines of therapy. 2. Male or Female subjects aged 18-70 years (at the time of signing the informed consent form).

  3. CD19 antigen expression of ≥20% (for B-ALL) or presence of CD19 expressing tumor cell population (for lymphoma).

  4. ECOG 0-2 points. 5. Life expectancy of at least 12 weeks. 6. Absolute CD3+ lymphocyte count in peripheral blood greater than 0.1*10^9 cells/L.

  7. Preserved organ function, defined as:
* Lung function: absence of hypoxemia according to pulse oximetry (SrO2 >91%) when breathing atmospheric air;
* Renal function: creatinine <130 µmol/L or ICF >60 ml/min per 1.73m2;
* Liver function: total bilirubin concentration less than 34 μmol/L, ALT concentration not exceeding more than 5 times the upper limit of reference values (except for Gilbert's syndrome);
* Cardiac function: stable hemodynamics and ejection fraction not less than 45%, absence of ejection in the pericardial cavity.

  8. Male or female patients with a very low probability of conception characterized by meeting at least one of the following criteria:
* Patient is not of reproductive potential. A female patient of no reproductive potential characterized by one of two criteria: (1) attainment of natural menopause (defined as 12 months of spontaneous amenorrhea in women >45 years of age or 6 months of spontaneous amenorrhea with a serum FSH concentration characteristic of the postmenopausal range as determined by the laboratory) or (2) bilateral ovariectomy and/or hysterectomy or bilateral fallopian tube ligation at least 6 weeks before screening.
* The patient is of reproductive potential and agrees to abstain from sexual activity or to use (including partner use) an acceptable method of contraception for the planned duration of the study. Acceptable contraceptive methods are hormonal contraception, intrauterine contraceptive device (IUD), diaphragm with spermicide, contraceptive sponge, condom, and vasectomy (performed at least 6 weeks prior to screening).

  9. Consent for continued follow-up for 15 years from study inclusion. 10. Adequate central or peripheral vascular access for the apheresis procedure. 11. The patient understands the study procedures, available alternative therapies, and study risks and voluntarily agrees to participate by providing written informed consent.

Exclusion Criteria:

1. Tumor cell surface CD19 expression level <20% for B-ALL by flow cytometry or no CD19 expression for lymphoma by immunohistochemical analysis.
2. Acute/active hepatitis B, C, or acute HIV infection, COVID-19.
3. Uncontrolled life-threatening infection (positive blood culture within 72 h prior to CAR-T product transfusion). Urinary tract infection is allowed. Patients receiving intravenous antibiotics prior to transfusion or in whom intravenous antibiotics have not been discontinued 7 days before inclusion in the study are not included. Prophylactic use of antibiotics, antiviral, and antifungal agents is allowed.
4. CD3+ T-lymphocyte content in peripheral blood is less than 0.1*10^9 cells/L.
5. Previous treatment with gene therapy products.
6. Clinically significant CNS pathology (epilepsy, generalized convulsive disorder, paresis, aphasia, stroke, severe brain damage, dementia, Parkinson's disease, cerebellar disease, organic cerebral syndrome, psychosis) at present or in the anamnesis.
7. NYHA class III or IV heart failure, coronary angioplasty or stenting, myocardial infarction, unstable angina, or any other significant cardiac pathology within the previous 6 months.
8. Associated genetic syndromes (such as Nijmegen syndrome, Kostman syndrome, Schwachman syndrome, or any other known bone marrow failure syndrome).
9. Pregnancy, planning pregnancy during the study, or lactation period.
10. Use of drugs or therapeutic interventions prohibited by the protocol (glucocorticosteroids, allogeneic cell therapy, GvHD therapy, chemotherapy, alemtuzumab, clofarabine, cladribine, mouse-derived biologics).
11. Participation in a clinical trial taking any investigational drug within 30 days prior to screening with the exception of investigational antimicrobials (antibiotics, antimycotics, and antivirals).
12. Any clinically relevant data that, in the opinion of the investigator, affects the patient's ability to enter the study and puts the patient at risk if they participate in the study.
13. Uncontrolled medical, psychological, familial, sociological, or geographical conditions and conditions that, in the investigator's opinion, make it impossible to achieve acceptable adherence to the study protocol and the subjects' unwillingness or inability to follow the protocol procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28 days
  Frequency of any adverse events (AEs) reported during the study period and AE characterization (severity, seriousness, etc.) on day 28
Primary Efficacy Outcome: ORR | 28 days
  Overall response rate (ORR) defined as the proportion of subjects with complete response (CR) or partial response (PR) on Day 28.

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Hematology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Offical approval of the trial by the Ministry of Health of the Russian Federation — https://grls.rosminzdrav.ru/CIPermissionMini.aspx?CIStatementGUID=4e10159b-46f4-4a5e-99cc-6209ec3cb388&CIPermGUID=6cee900a-c359-4873-8b17-a506839f0acd